CLINICAL TRIAL: NCT02324569
Title: A Phase 4, Multicenter, Randomized, Double-blind, Placebo-controlled, Parallel-group, Comparative Study and a Phase 4, Multicenter, Open-label, Long-term Study to Evaluate the Safety and Efficacy of SYR-472 When Orally Administered at a Dose of 100 mg Once Weekly as an add-on to Insulin Therapy in Patients With Type 2 Diabetes Mellitus and Inadequate Glycemic Control Despite Treatment With Insulin Preparations in Addition to Diet and/or Exercise Therapy
Brief Title: A Phase 4, Randomized, Double-blind, Parallel-group, Comparative Study and a Phase 4, Open-label, Long-term Study of SYR-472 (100 mg) in Combination With Insulin in Patients With Type 2 Diabetes
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SYR-472/CCT-101; U1111-1164-8291 (Other: WHO)
Record Dates: First submitted 2014-12-19; First posted 2014-12-24 (Estimated); Results first posted 2019-02-11 (Actual); Last update posted 2023-12-12 (Actual); Status verified 2023-12

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Pharmacological therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — trelagliptin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment Group I (Experimental): One tablet of SYR-472 100 mg orally once weekly before breakfast
  Interventions: Drug: SYR-472
- Treatment Group II (Experimental): One tablet of SYR-472 100 mg orally or one placebo tablet orally once weekly before breakfast
  Interventions: Drug: SYR-472; Drug: Placebo

INTERVENTIONS:
Drug: SYR-472 — SYR-472 tablets
Drug: Placebo — Placebo tablets
  Arms: Treatment Group II

SUMMARY:
The purposes of this study is to evaluate the efficacy and safety of SYR-472 when administered at a dose of 100 mg once weekly as an add-on to insulin therapy compared with placebo in patients with type 2 diabetes mellitus and inadequate glycemic control despite treatment with insulin preparations in addition to diet and/or exercise therapy; and to evaluate the long-term efficacy and safety of SYR-472 when administered at a dose of 100 mg once weekly as an add-on to insulin therapy in patients with type 2 diabetes mellitus and inadequate glycemic control despite treatment with insulin preparations in addition to diet and/or exercise therapy.

DETAILED DESCRIPTION:
This is a phase 4, multicenter, randomized, double-blind, parallel-group, comparative study using placebo (Treatment Period I) and a phase 4, multicenter, open-label, long-term study (Treatment Period II) to evaluate the efficacy and safety of SYR-472 when administered at a dose of 100 mg as an add-on to insulin therapy in patients with type 2 diabetes mellitus and inadequate glycemic control despite treatment with insulin preparations in addition to diet and/or exercise therapy.

ELIGIBILITY:
Inclusion Criteria:

Participant eligibility is determined according to the following criteria:

1. The participant has a diagnosis of type 2 diabetes mellitus.
2. The participant has a fasting C-peptide level of 0.6 ng/mL or higher at the start of the screening period (Week -6) and Week -2 of the screening period.
3. The participant has a Haemoglobin A1c (HbA1c) value of 7.5% or higher but less than 10.0% at Week -2 of the screening period.
4. The participant has an HbA1c value difference between the start of the screening period (Week -6) and Week -2 of the screening period within 10.0%* (* rounded to one decimal place) of the HbA1c value at the start of the screening period (Week -6).
5. The participant has been on a fixed diet and/or exercise therapy (if any) from at least 6 weeks prior to the start of the screening period (Week -6).
6. The participant is being treated with insulin preparations alone (≥8 units/day and ≤40 units/day) ** from at least 6 weeks prior to the start of the screening period (Week -6) at a fixed dose and regimen of the insulin preparation.

   * The participant on any one of the following insulin monotherapies: mixed (rapid-acting or short-acting insulin containing no more than 30% volume), intermediate-acting, or long-acting soluble insulin preparations
7. The participant is deemed appropriate for treatment with a combination of insulin and another antidiabetic drug at the start of the screening period (Week -6) by the investigator or subinvestigator.
8. The participants with controlled and stable blood pressure will not need any change in the dose of antihypertensive drugs (including discontinuation and suspension) or additional antihypertensive drugs during the study period as assessed by the investigator or subinvestigator.
9. The participant is male or female and aged 20 years or older at the time of informed consent.
10. A female participant of childbearing potential who is sexually active with a nonsterilized male partner agrees to use routinely adequate contraception from signing of informed consent until one month after the end of the study.
11. In the opinion of the investigator or subinvestigator, the participant is capable of understanding and complying with protocol requirements.
12. The participant signs and dates a written, informed consent form prior to the initiation of any study procedures.

Exclusion Criteria:

Any participant who meets any of the following criteria will not qualify for entry into the study:

1. The participants has clinical manifestations of hepatic impairment [e.g., Aspartate Aminotransferase (AST) or Alanine Aminotransferase (ALT) ≥2.5 times the upper limit of normal or total bilirubin of ≥2.0 mg/dL at the start of the screening period (Week -6) or at Week -2 of the screening period].
2. The participant has moderate or severe renal impairment or end-stage renal failure [e.g., creatinine clearance (Ccr) <50 mL/min at the start of the screening period (Week -6) or Week -2 of the screening period].
3. The participant has any serious cardiac diseases, cerebrovascular disorders, or serious pancreatic or hematological diseases (e.g., participants who require inpatient treatment or are hospitalized for treatment within 24 weeks prior to the start of the screening period).
4. The participant has, in the judgment of the investigator or subinvestigator, clinically significant abnormal hematological parameters of hemoglobin, hematocrit, or erythrocytes at the start of the screening period (Week - 6) or Week -2 of the screening period.
5. The participant has a systolic blood pressure of 180 mmHg or higher or a diastolic blood pressure of 110 mmHg or higher during the screening period.
6. The participant is on at least two antidiabetic therapies other than one insulin preparation one day before 6 weeks prior to the start of the screening period (Week -6) (43 days prior to the start of the screening period).
7. The participants altered the dose and regimen of their insulin preparation within 6 weeks prior to the start of the screening period or during the screening period.
8. The participant experienced hypoglycemia (participants with a blood glucose level of ≤70 mg/dL or hypoglycemic symptoms) within 6 weeks prior to the start of the screening period or during the screening period (at least twice per week).
9. The participant has a fasting blood glucose level of 240 mg/dL or higher at the start of the screening period (Week -6) or at Week -2 of the screening period.
10. The participant has malignancies.
11. The participant has a history of hypersensitivity or allergies to dipeptidyl peptidase 4 (DPP-4) inhibitors or insulin preparations.
12. The participant has a history of gastrectomy or small intestinal resection.
13. The participant is habitual drinker consuming a daily average of more than 100 mL of alcohol.
14. The participant has a history of drug abuse (defined as the use of an illegal drug) or alcohol dependence.
15. The participant is required to take excluded medications during the study period.
16. The participant has received SYR-472 in a previous clinical study.
17. The participant is deemed to be in a condition contraindicating treatment as specified in the package insert of insulin preparations by the investigator or subinvestigator.
18. The participant received any investigational products (including study drugs in a post-marketing clinical study) within 12 weeks prior to the start of the screening period.
19. The participant is participating in other clinical studies at the time of informed consent.
20. If female, the participant is pregnant or lactating or intending to become pregnant before, during, or within 1 month after participating in this study; or intending to donate ova during such time period.
21. The participant is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
22. The participant is hospitalized during the screening period or deemed as requiring hospitalization during the study period by the investigator or subinvestigator, unless the hospitalization is for short-term evaluations including complete health checkups.
23. The participant is deemed to be ineligible for the study for any other reason by the investigator or subinvestigator.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2014-12-27 (Actual); Primary Completion 2016-12-28 (Actual); Study Completion 2016-12-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (65):
- Japan (65):
  - Nagoya, Aichi-ken
  - Hirosaki, Aomori
  - Kurume, Fukuoka
  - Sapporo, Hokkaido
  - Koga, Ibaragi
  - Mito, Ibaragi
  - Naka, Ibaragi
  - Tsuchiura, Ibaragi
  - Ushiku, Ibaragi
  - Kanazawa, Ishikawa-ken
  - Satsumakawauchi, Kagoshima-ken
  - Chigasaki, Kanagawa
  - Fujisawa, Kanagawa
  - Sendai, Miyagi
  - Hirakata, Osaka
  - Kashihara, Osaka
  - Suita, Osaka
  - Ageo, Saitama
  - Sangou, Saitama
  - Hamamatsu, Shizuoka
  - Shimada, Shizuoka
  - Koyama, Tochigi
  - Shimono, Tochigi
  - Chiyoda-ku, Tokyo
  - Nerima-ku, Tokyo
  - Shinjuku-ku, Tokyo
  - Suginami-ku, Tokyo
  - Tama, Tokyo
  - Shimonoseki, Yamaguchi
  - Shunann, Yamaguchi
  - Ageo
  - Aomori
  - Chiba
  - Chigasaki
  - Chiyoda-ku
  - Fujisawa
  - Fukuoka
  - Hamamatsu
  - Hirakata
  - Hirosaki
  - Kagoshima
  - Kanazawa
  - Kashiwara
  - Koga
  - Koyama
  - Kumamoto
  - Kurume
  - Kyoto
  - Mito
  - Nagoya
  - Naka
  - Nerima-ku
  - Osaka
  - Sangō
  - Satsumakawauchi
  - Sendai
  - Shimada
  - Shimono
  - Shimonoseki
  - Shinjuku-ku
  - Shizuoka
  - Suginami-ku
  - Tama
  - Toyama
  - Tsuchiura

IPD SHARING:
Plan to Share IPD: Yes

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 43 investigative sites in Japan, from 27 December 2014 to 28 December 2016.
Pre-assignment Details: Participants with a historical diagnosis of type 2 diabetes mellitus with inadequate glycemic control despite treatment with insulin therapy were enrolled in 1 of the 2 groups: Group I: 100 milligram (mg) SYR-472 in Period I followed by 100 mg SYR-472 in Period II, Group II: SYR-472 Placebo in Period I followed by 100 mg SYR-472 in Period II.
Groups:
- Treatment Group I: SYR-472 100 mg, one tablet, orally before breakfast, weekly for up to Week 12 as Period I, followed by SYR-472 100 mg, one tablet, orally before breakfast, weekly for up to Week 52 as Period II of this study. Participants treated with insulin therapy throughout study.
- Treatment Group II: SYR-472 placebo, one tablet, orally before breakfast, weekly for up to Week 12 as Period I, followed by SYR-472 100 mg, one tablet, orally before breakfast, weekly for up to Week 52 as Period II of this study. Participants treated with insulin therapy throughout study.
Period: Overall Study
Arm/Group | Treatment Group I | Treatment Group II
Started | 116 | 124
Completed | 100 | 103
Not Completed | 16 | 21
Not completed — Pretreatment Event/Adverse Event | 9 | 10
Not completed — Voluntary Withdrawal | 3 | 6
Not completed — Lack of Efficacy | 2 | 3
Not completed — Change Insulin Dosage Exceeding Criteria | 0 | 2
Not completed — Inconvenient Schedule | 2 | 0

BASELINE CHARACTERISTICS:
Population: Randomized set: Randomized set included all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group I | Treatment Group II | Total
Number analyzed (Participants) | 116 | 124 | 240
Age, Continuous [Mean (Standard Deviation); unit: Years] | 57.9 (10.89) | 58.5 (11.11) | 58.2 (10.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 42 | 68
  Male | 90 | 82 | 172
Region of Enrollment [Number; unit: Participants] — All participants were enrolled in Japan.
  Participants
    Japan | 116 | 124 | 240
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index = weight (kg)/[height (m)^2]
  kg/m^2 | 25.39 (3.593) | 25.16 (3.402) | 25.27 (3.490)
Duration of Diabetes [Mean (Standard Deviation); unit: Months] — Mean duration between start of study and first time of diagnosis of type 2 diabetes mellitus was reported.
  Months | 125.9 (92.75) | 143.6 (90.23) | 135.0 (91.69)
Type of Insulin Preparation [Count of Participants; unit: Participants]
  Pre-Mixed | 48 | 47 | 95
  Intermediate-Acting | 3 | 9 | 12
  Long-Acting | 65 | 68 | 133
Daily Dose of Insulin Preparation at Week -6 [Mean (Standard Deviation); unit: Unit] | 19.8 (9.32) | 18.8 (8.88) | 19.3 (9.09)
Creatinine Clearance (Ccr) [Mean (Standard Deviation); unit: Milliliter (mL)/minute (min)] | 109.3 (36.09) | 107.4 (40.28) | 108.3 (38.24)
Haemoglobin A1c (HbA1c) [Mean (Standard Deviation); unit: Percent] | 8.42 (0.677) | 8.50 (0.675) | 8.46 (0.675)
Fasting Plasma Glucose [Mean (Standard Deviation); unit: Milligram (mg)/ Deciliter (dL)] | 160.6 (32.86) | 167.3 (34.02) | 164.1 (33.56)
2-hour (hr) Postprandial Plasma Glucose [Mean (Standard Deviation); unit: mg/dL] | 290.0 (52.08) | 286.1 (54.03) | 288.0 (52.97)
Fasting C-Peptide [Mean (Standard Deviation); unit: Nanogram (ng)/mL] | 1.07 (0.527) | 1.16 (0.647) | 1.12 (0.593)
Glycoalbumin [Mean (Standard Deviation); unit: Percent] | 23.53 (3.343) | 23.70 (3.290) | 23.62 (3.310)
1,5-Anhydroglucitol [Mean (Standard Deviation); unit: Microgram (μg)/mL] | 3.39 (2.349) | 3.28 (2.978) | 3.33 (2.688)
Insulinogenic Index [Mean (Standard Deviation); unit: microunits*dL/mg*mL] — Insulinogenic Index=Increment of insulin at 30 minutes post-meal / Increment of blood glucose at 30 minutes post-meal
  microunits*dL/mg*mL | 0.29 (0.279) | 0.38 (0.687) | 0.34 (0.525)

OUTCOME MEASURES:

1. Primary Outcome: Change in HbA1c From Baseline at the End of Treatment Period I (End of Treatment Period I - End of the Screening Period)
Time Frame: End of the screening period (Week 0) and End of Treatment Period I (Up to Week 12)
Population: Full Analysis Set: All randomized participants who received at least one dose of study drug.
Measure: Least Squares Mean (Standard Error); unit: Percent
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
Percent | -0.56 (0.070) | 0.07 (0.067)
Statistical Analysis 1: Comparison: Treatment Group I vs Treatment Group II; Test type: Superiority; p < 0.0001, ANCOVA; Least square (LS) mean difference = -0.63, 95% CI 2-sided [-0.826 to -0.443], Standard Error of Mean 0.097

2. Primary Outcome: Number of Participants Reporting One or More Treatment-Emergent Adverse Events (TEAEs) That Occurred Before Start of Treatment Period II
Description: Reported data is the number of participants reporting one or more TEAEs that occurred before start of Treatment Period II in Treatment Group I and Treatment Group II.
Time Frame: Up to Week 12
Population: Safety Analysis Set: The safety analysis set was defined as the participants who received at least 1 dose of the study drug for the treatment period.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
Participants | 51 | 59

3. Secondary Outcome: Change From Baseline in HbA1c
Description: Reported data was the change from baseline in HbA1c at each time point.
Time Frame: Baseline and Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, End of Treatment Period I (Up to Week 12) and End of Treatment Period II (Up to Week 52)
Population: Full Analysis Set: All randomized participants who received at least one dose of study drug. The analyzed numbers for each arm were participants who were evaluable for this outcome measure at the given time point.
Measure: Mean (Standard Deviation); unit: Percent
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
Percent
  Week 2: number analyzed (Participants) | 115 | 124
  Week 2 | -0.16 (0.240) | 0.01 (0.229)
  Week 4: number analyzed (Participants) | 113 | 124
  Week 4 | -0.38 (0.327) | -0.06 (0.396)
  Week 8: number analyzed (Participants) | 113 | 123
  Week 8 | -0.50 (0.573) | -0.04 (0.612)
  Week 12: number analyzed (Participants) | 111 | 120
  Week 12 | -0.55 (0.708) | 0.08 (0.793)
  Week 16: number analyzed (Participants) | 112 | 117
  Week 16 | -0.51 (0.793) | -0.16 (0.840)
  Week 20: number analyzed (Participants) | 111 | 113
  Week 20 | -0.42 (0.836) | -0.41 (0.797)
  Week 24: number analyzed (Participants) | 109 | 112
  Week 24 | -0.38 (0.864) | -0.49 (0.812)
  Week 28: number analyzed (Participants) | 107 | 111
  Week 28 | -0.42 (0.884) | -0.55 (0.832)
  Week 32: number analyzed (Participants) | 107 | 109
  Week 32 | -0.41 (0.872) | -0.57 (0.791)
  Week 36: number analyzed (Participants) | 105 | 106
  Week 36 | -0.42 (0.817) | -0.58 (0.740)
  Week 40: number analyzed (Participants) | 103 | 105
  Week 40 | -0.35 (0.884) | -0.62 (0.779)
  Week 44: number analyzed (Participants) | 102 | 103
  Week 44 | -0.34 (0.895) | -0.67 (0.772)
  Week 48: number analyzed (Participants) | 100 | 103
  Week 48 | -0.44 (0.804) | -0.69 (0.794)
  Week 52: number analyzed (Participants) | 99 | 102
  Week 52 | -0.48 (0.799) | -0.70 (0.711)
  End of Treatment Period I: number analyzed (Participants) | 115 | 124
  End of Treatment Period I | -0.56 (0.710) | 0.07 (0.788)
  End of Treatment Period II: number analyzed (Participants) | 115 | 118
  End of Treatment Period II | -0.43 (0.827) | -0.60 (0.831)

4. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose
Description: Reported data was the change from baseline in fasting plasma glucose at each time point.
Time Frame: Baseline and Week 2, 4, 8, 12, 16, 20, 24, 28, 32, 36, 40, 44, 48, 52, 53, End of Treatment Period I (Up to Week 12) and End of Treatment Period II (Up to Week 52)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
mg/dL
  Week 2: number analyzed (Participants) | 115 | 124
  Week 2 | -10.3 (29.73) | 0.1 (28.98)
  Week 4: number analyzed (Participants) | 113 | 124
  Week 4 | -12.6 (32.19) | -4.0 (36.49)
  Week 8: number analyzed (Participants) | 113 | 123
  Week 8 | -9.3 (32.13) | -0.9 (39.37)
  Week 12: number analyzed (Participants) | 111 | 120
  Week 12 | -2.0 (39.65) | 2.0 (42.04)
  Week 16: number analyzed (Participants) | 112 | 117
  Week 16 | -1.4 (41.31) | -9.0 (37.24)
  Week 20: number analyzed (Participants) | 111 | 113
  Week 20 | -3.1 (39.65) | -10.4 (38.68)
  Week 24: number analyzed (Participants) | 109 | 112
  Week 24 | -3.0 (36.08) | -10.3 (39.79)
  Week 28: number analyzed (Participants) | 107 | 111
  Week 28 | -4.5 (38.76) | -10.5 (37.50)
  Week 32: number analyzed (Participants) | 107 | 109
  Week 32 | -6.9 (39.46) | -12.9 (35.75)
  Week 36: number analyzed (Participants) | 105 | 106
  Week 36 | -6.0 (35.58) | -14.9 (33.97)
  Week 40: number analyzed (Participants) | 104 | 105
  Week 40 | -3.7 (40.45) | -14.7 (36.34)
  Week 44: number analyzed (Participants) | 102 | 103
  Week 44 | -4.9 (36.88) | -18.0 (38.43)
  Week 48: number analyzed (Participants) | 100 | 103
  Week 48 | -8.8 (38.00) | -19.8 (35.38)
  Week 52: number analyzed (Participants) | 99 | 102
  Week 52 | -10.0 (43.40) | -21.0 (33.99)
  Week 53: number analyzed (Participants) | 105 | 113
  Week 53 | -1.3 (45.44) | -13.2 (34.49)
  End of Treatment Period I: number analyzed (Participants) | 115 | 124
  End of Treatment Period I | -2.8 (39.40) | 0.8 (42.44)
  End of Treatment Period II: number analyzed (Participants) | 115 | 118
  End of Treatment Period II | -8.1 (42.48) | -18.3 (35.81)

5. Secondary Outcome: Change From Baseline in Plasma Glucose Measured by the Meal Tolerance Test in Treatment Period I
Description: Reported data was the change from pre-meal in plasma glucose measured by the meal tolerance test at each time point.
Time Frame: Pre-meal and 0.5, 1, and 2 hr after-meal at Week 0 and 0.5, 1, and 2 hr after-meal at the End of Treatment Period I (Up to Week 12)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
mg/dL
  Pre-meal at the End of Treatment Period I: number analyzed (Participants) | 77 | 84
  Pre-meal at the End of Treatment Period I | -9.5 (34.13) | 0.5 (45.17)
  0.5 hr at the End of Treatment Period I: number analyzed (Participants) | 77 | 84
  0.5 hr at the End of Treatment Period I | -17.6 (36.82) | 3.5 (51.12)
  1 hr at the End of Treatment Period I: number analyzed (Participants) | 77 | 84
  1 hr at the End of Treatment Period I | -28.6 (43.08) | -1.2 (51.02)
  2 hr at the End of Treatment Period I: number analyzed (Participants) | 77 | 84
  2 hr at the End of Treatment Period I | -29.9 (42.23) | 2.3 (59.89)

6. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Vital Signs Before Start of Treatment Period II
Description: Here "mmHg" is Millimeter of mercury.
Time Frame: Up to Week 12
Population: Safety Analysis Set: The safety analysis set was defined as the participants who received at least 1 dose of the study drug for the treatment period. The analyzed numbers for each arm were participants who were evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
Participants
  Diastolic Blood Pressure <50 mmHg: number analyzed (Participants) | 115 | 124
  Diastolic Blood Pressure <50 mmHg | 1 | 1
  Pulse <50 Beats per minute(bpm): number analyzed (Participants) | 115 | 124
  Pulse <50 Beats per minute(bpm) | 1 | 2

7. Secondary Outcome: Number of Participants With Markedly Abnormal Values of ECG Parameters Before Start of Treatment Period II
Description: Here "QTcF" is Corrected QT interval by Fridericia formula, and "msec" is millisecond.
Time Frame: Up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
Participants
  QTcF Interval >450 msec: number analyzed (Participants) | 113 | 122
  QTcF Interval >450 msec | 2 | 4
  Change from Baseline in QTcF Interval >30 msec: number analyzed (Participants) | 113 | 122
  Change from Baseline in QTcF Interval >30 msec | 2 | 1

8. Secondary Outcome: Number of Participants With Markedly Abnormal Values of Laboratory Parameters (Total Bilirubin >2.0) Before Start of Treatment Period II
Time Frame: Up to Week 12
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
Participants | 1 | 1

9. Secondary Outcome: Number of Participants With Total Hypoglycaemia After 1st Dose of Study Drug and Before Start of Treatment Period II
Time Frame: Up to Week 53
Population: as for outcome 6
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
Participants | 17 | 16

10. Secondary Outcome: Change From Baseline in Self-Monitoring of Blood Glucose Before Breakfast
Description: Reported data was the change from baseline in self-monitoring of blood glucose before breakfast.
Time Frame: Baseline and Day 2, 3, 4, 5, 6, 7, and 8 in each Treatment Period (I and II) (Totally up to Week 17)
Population: Safety Analysis Set: The safety analysis set was defined as the participants who received at least 1 dose of the study drug for the treatment period. The analyzed numbers for each arm were participants who were evaluable for this outcome measure at the given time point.
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Treatment Group I | Treatment Group II
Number analyzed (Participants) | 116 | 124
mg/dL
  Day 2 on Treatment Period I: number analyzed (Participants) | 110 | 115
  Day 2 on Treatment Period I | 9.7 (41.21) | 5.6 (39.02)
  Day 3 on Treatment Period I: number analyzed (Participants) | 108 | 114
  Day 3 on Treatment Period I | 4.3 (35.22) | -0.9 (41.35)
  Day 4 on Treatment Period I: number analyzed (Participants) | 108 | 112
  Day 4 on Treatment Period I | 1.6 (43.99) | -3.0 (41.55)
  Day 5 on Treatment Period I: number analyzed (Participants) | 109 | 113
  Day 5 on Treatment Period I | -6.7 (41.51) | -0.9 (38.22)
  Day 6 on Treatment Period I: number analyzed (Participants) | 108 | 115
  Day 6 on Treatment Period I | -7.0 (33.79) | 2.2 (43.78)
  Day 7 on Treatment Period I: number analyzed (Participants) | 109 | 113
  Day 7 on Treatment Period I | -0.2 (38.15) | -0.3 (37.55)
  Day 8 on Treatment Period I: number analyzed (Participants) | 110 | 113
  Day 8 on Treatment Period I | -3.8 (39.63) | 2.0 (37.70)
  Day 2 on Treatment Period II: number analyzed (Participants) | 105 | 109
  Day 2 on Treatment Period II | -6.8 (41.98) | 7.1 (51.90)
  Day 3 on Treatment Period II: number analyzed (Participants) | 104 | 111
  Day 3 on Treatment Period II | -10.2 (39.95) | 5.8 (44.25)
  Day 4 on Treatment Period II: number analyzed (Participants) | 107 | 112
  Day 4 on Treatment Period II | -5.7 (45.52) | -1.7 (49.40)
  Day 5 on Treatment Period II: number analyzed (Participants) | 106 | 106
  Day 5 on Treatment Period II | -5.2 (41.24) | -2.8 (47.25)
  Day 6 on Treatment Period II: number analyzed (Participants) | 106 | 107
  Day 6 on Treatment Period II | -8.5 (39.04) | -3.4 (40.67)
  Day 7 on Treatment Period II: number analyzed (Participants) | 105 | 107
  Day 7 on Treatment Period II | -7.7 (35.93) | -4.9 (44.21)
  Day 8 on Treatment Period II: number analyzed (Participants) | 106 | 107
  Day 8 on Treatment Period II | -9.4 (35.91) | -7.8 (43.85)

ADVERSE EVENTS:
Time Frame: Baseline up to Week 53
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment. On serious adverse events table, only events that occurred after 1st dose of SYR-472 were reported.
Arm/Group | Treatment Group I | Treatment Group II
Serious Adverse Events (participants affected / at risk) | 16/116 | 9/119
Other Adverse Events (participants affected / at risk) | 59/116 | 54/119
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group I (N=116) | Treatment Group II (N=119)
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Cardiac failure congestive (Cardiac disorders) | 1 | 0
Coronary artery aneurysm (Cardiac disorders) | 0 | 1
Coronary artery stenosis (Cardiac disorders) | 0 | 1
Mitral valve incompetence (Cardiac disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 2 | 1
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0
Enteritis (Gastrointestinal disorders) | 1 | 0
Ileus paralytic (Gastrointestinal disorders) | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 1
Pancreatolithiasis (Gastrointestinal disorders) | 0 | 1
Accident (Injury, poisoning and procedural complications) | 1 | 0
Arterial injury (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 1 | 0
Muscle rupture (Injury, poisoning and procedural complications) | 1 | 0
Radial nerve injury (Injury, poisoning and procedural complications) | 1 | 0
Spinal cord injury cervical (Injury, poisoning and procedural complications) | 1 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Medullary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Renal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basilar artery stenosis (Nervous system disorders) | 0 | 1
Cerebellar infarction (Nervous system disorders) | 0 | 1
Loss of consciousness (Nervous system disorders) | 0 | 1
Completed suicide (Psychiatric disorders) | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Cerebral Infarction (Nervous system disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Group I (N=116) | Treatment Group II (N=119)
Dental caries (Gastrointestinal disorders) | 7 | 1
Nasopharyngitis (Infections and infestations) | 40 | 31
Hypoglycaemia (Metabolism and nutrition disorders) | 22 | 18
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 8
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 7 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.